CLINICAL TRIAL: NCT04693676
Title: A Phase 1 Study Evaluating Safety and Efficacy of C-CAR039 Treatment in Subjects With Relapsed and/or Refractory NHL
Brief Title: A Study of C-CAR039 Treatment in Subjects With r/r NHL Subjects Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0702-025
Record Dates: First submitted 2020-12-03; First posted 2021-01-05 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-05

CONDITIONS: Non-Hodgkin's B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prizloncabtagene autoleucel (Experimental): Prizlon-cel will be intravenously administered as a single infusion after lymphodepletion
  Interventions: Biological: Prizloncabtagene Autoleucel

INTERVENTIONS:
Biological: Prizloncabtagene Autoleucel — Autologous 2nd generation CD19/CD20-directed CAR-T cells, single infusion intravenously
  Other Names: C-CAR039

SUMMARY:
This is a single-arm, open label, dose escalation, phase I study of C-CAR039 in adults with relapsed/refractory B-cell Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
This is a single-arm, open label, "3+3" dose escalation, phase I study to evaluate the safety and preliminary efficacy of C-CAR039 in adults with relapsed/refractory B-cell Non-Hodgkin's Lymphoma. 10 patients are planned to be enrolled.

Following consent, enrolled subjects will undergo a leukapheresis procedure to collect autologous mononuclear cells for manufacture of C-CAR039. Following manufacture of the drug product, subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide prior to C-CAR039 infusion. All subjects who have received C-CAR039 infusion will be followed for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteered to participate in the study and signed the Informed Consent;
2. Age between 18 and 70 (including 18 and 70), male or female;
3. Expected survival ≥ 12 weeks;
4. ECOG score 0-2
5. CD19 or CD20 positive B-NHL confirmed by cytology or histology according to WHO2016 criteria, including DLBCL, PMBCL, tFL, FL and MCL;
6. Relapsed or refractory disease after ≥ 2 lines (for FL, at least 3 lines) of standard therapy or relapsed after autologous stem cell transplantation (ASCT)
7. For CD20-positive subjects, they should have received at least one regimen containing anti-CD20-targeted therapy (such as rituximab). If they do not complete the regimen due to intolerance, the cause of intolerance should be recorded;
8. No contraindications of apheresis;
9. At least one measurable lesion according to Lugano 2014 criteria;
10. Adequate organ function.

Exclusion Criteria:

1. Malignant tumors other than B-NHL within 5 years prior to screening, except cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and breast ductal carcinoma in situ after radical surgery;
2. Active HIV, HBV, HCV or treponema pallidum infection ;
3. Any instability of systemic disease, including but not limited to active infection (except local infection), severe cardiac, liver, kidney, or metabolic disease need therapy;
4. Any uncontrolled, active disease that prevents participation in the trial;
5. Female subjects who have been pregnant or breastfeeding, or who plan to conceive during or within 1 year after treatment, or male subjects' partner plans to conceive within 1 year after their cell transfusion;
6. Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment;
7. Patients who have been previously infected with tuberculosis;
8. Administered Corticosteroids and/or other immunosuppressants within 7 days before apheresis. and 5 days before the infusion of C-CAR039;
9. Patients with central nervous system involvement;
10. Any systemic antitumor therapy was performed within 2 weeks before conditional treatment chemotherapy pretreatment;
11. Any situation that the investigator believes would compromise the safety of the subject or interfere with the purpose of the study;
12. Those with medical conditions that prevent them from signing the written informed consent or from complying with the study procedures; or those who are unwilling or unable to comply with the study requirements.
13. Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
MTD | Up to 24 months after C-CAR039 infusion
  maximum tolerated dose or clinical recommended dose
DLT | Up to 28 days after C-CAR039 infusion
  Dose limiting toxicity
AE/SAE/AESI | Up to 24 months after C-CAR039 infusion
  adverse events (AE), serious adverse event (SAE), adverse events of sepical interest (AESI) (including cytokine release syndrome (CRS), and nerve toxicity), laboratory tests (type, frequency and severity), vital signs and ECG abnormality rate.

SECONDARY OUTCOMES:
C-CAR039 CAR expansion and persistence | Up to 24 Months after C-CAR039 infusion
  After C-CAR039 infusion, peripheral blood EXP039 CAR expansion and persistence in vivo, including Cmax, Tmax, AUC0-28day, Tlast
Overall response rate (ORR) | Up to 24 Months after C-CAR039 infusion
  Complete response (CR) rate plus partial response (PR) rate by Lugano 2014 criteria
Duration of response (DOR) | Up to 24 Months after C-CAR039 infusion
  The time from the date of first response (PR or better) to the date of disease progression or death after C-CAR039 infusion
Progression-free survival (PFS) | Up to 24 Months after C-CAR039 infusion
  The time from C-CAR039 infusion to the date of progression as assessed by Lugano 2014 criteria or death
Overall survival (OS) | Up to 24 Months after C-CAR039 infusion
  The time from C-CAR039 infusion to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, PhD&MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu W, Li P, Zhou L, Yang M, Ye S, Zhu D, Huang J, Yao X, Zhang Y, Li L, Zhao J, Zhu K, Li J, Zheng C, Lan L, Wan H, Yao Y, Zhang H, Zhou D, Jin J, Liang A. A phase 1 trial of prizloncabtagene autoleucel, a CD19/CD20 CAR T-cell therapy for relapsed/refractory B-cell non-Hodgkin lymphoma. Blood. 2025 Apr 3;145(14):1526-1535. doi: 10.1182/blood.2024026401. PMID 39813680